CLINICAL TRIAL: NCT00316927
Title: A Randomized Phase III Trial of Dexamethasone and Aspirin (DA) Versus Dexamethasone, Diethylstilbestrol and Aspirin (DAS) in Locally Advanced or Metastatic Cancer of the Prostate - Immediate Versus Deferred Diethylstilbestrol
Brief Title: Dexamethasone, Aspirin, and Diethylstilbestrol in Treating Patients With Locally Advanced or Metastatic Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Bartholomew's Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: BARTS-DAVDAS; CDR0000472404 (Registry Identifier: PDQ (Physician Data Query)); EU-20610; ISRCTN13255144
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2007-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Aspirin; Dexamethasone; Diethylstilbestrol

INTERVENTIONS:
Drug: acetylsalicylic acid
Drug: dexamethasone
Drug: diethylstilbestrol

SUMMARY:
RATIONALE: Giving dexamethasone together with aspirin and diethylstilbestrol may be effective in lowering prostate-specific antigen levels and may slow or stop the growth of prostate cancer. It is not yet known which schedule of dexamethasone, aspirin, and diethylstilbestrol is more effective in treating prostate cancer.

PURPOSE: This randomized phase III trial is studying dexamethasone and aspirin when given together with two different schedules of diethylstilbestrol to compare how well they work in treating patients with locally advanced or metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the prostate-specific antigen (PSA) response in patients with locally advanced or metastatic prostate cancer treated with dexamethasone and aspirin with delayed vs immediate diethylstilbestrol.

Secondary

* Compare the overall response rate in patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.
* Compare the progression-free and overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are stratified according to ECOG performance status (0 vs 1-3), prostate-specific antigen (PSA) response to prior therapy (PSA normalization vs inability to normalize), and bone scan (positive vs negative for bony metastases). Patients are randomized to 1 of 2 treatment arms.

* Arm I (deferred diethylstilbestrol): Patients receive oral dexamethasone and oral acetylsalicyclic acid once daily (DA). Subsequent to treatment failure with DA, patients continue to receive DA as before in addition to oral diethylstilbestrol once daily (DAS). Treatment with DAS continues in the absence of disease progression or unacceptable toxicity.
* Arm II (immediate diethylstilbestrol): Patients receive oral dexamethasone, oral acetylsalicyclic acid, and oral diethylstilbestrol once daily (DAS). Treatment continues in the absence of disease progression or unacceptable toxicity.

Quality of life is evaluated monthly during study treatment.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 260 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of adenocarcinoma of the prostate

  * Elevated prostate-specific antigen (PSA)
* Failed previous treatments, including gonadatropan regulatory hormone analogue therapy, radiotherapy, surgery, or any combination of these
* Biochemically castrate (testosterone < 1 nmol/L) at baseline

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 3 months
* ECOG performance status 0-3
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count (neutrophils and bands) ≥ 2,000/mm^3
* Platelet count ≥ 50,000/mm^3
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST or ALT ≤ 3 times ULN
* Creatinine ≤ 1.5 times ULN
* Able to swallow tablets
* No other malignancy within the past 3 years except basal cell skin cancer
* No previous thromboembolic disease, including stroke, venous or arterial thrombosis, and myocardial infarction with ongoing angina pectoris

  * Prior uncomplicated myocardial infarction allowed
* No diabetes mellitus if treatment titration is thought to be difficult or inappropriate
* No active gastric or duodenal ulcer

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior concurrent bisphosphonates allowed
* No concurrent investigational agents or participation in another investigational drug study
* No other concurrent antineoplastic therapy, including new estrogen therapy, radiation therapy, or PC-SPES
* No other concurrent corticosteroids (e.g., dexamethasone for nausea or vomiting) except those prescribed in the study regimen

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2002-12; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Prostate-specific antigen (PSA) response

SECONDARY OUTCOMES:
Overall response
Quality of life
Progression-free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shamash, MD, FRCP, Study Chair — St. Bartholomew's Hospital
Locations (15):
- United Kingdom (15):
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Burnley General Hospital, Burnley, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Eastbourne District General Hospital, Eastbourne, England
  - Whipps Cross Hospital, London, England
  - Saint Bartholomew's Hospital, London, England
  - Chelsea Westminster Hospital, London, England
  - Maidstone Hospital, Maidstone, England
  - Milton Keynes General Hospital, Milton Keynes, England
  - Churchill Hospital, Oxford, England
  - Oldchurch Hospital, Romford, England
  - Torbay Hospital, Torquay Devon, England
  - Weston General Hospital, Weston-super-Mare, England
  - Worthing Hospital, Worthing, England
  - Cancer Care Centre at York Hospital, York, England

REFERENCES:
- [Result] Shamash J, Powles T, Sarker SJ, Protheroe A, Mithal N, Mills R, Beard R, Wilson P, Tranter N, O'Brien N, McFaul S, Oliver T. A multi-centre randomised phase III trial of Dexamethasone vs Dexamethasone and diethylstilbestrol in castration-resistant prostate cancer: immediate vs deferred Diethylstilbestrol. Br J Cancer. 2011 Feb 15;104(4):620-8. doi: 10.1038/bjc.2011.7. Epub 2011 Feb 1. PMID 21285990